CLINICAL TRIAL: NCT00799175
Title: Local Infiltration Analgesia With Ropivacaine, Ketorolac and Epinephrine Intra- and Postoperatively in Total Knee Arthroplasty
Brief Title: Local Infiltration Analgesia Following Total Knee Arthroplasty
Acronym: RAK-total
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Kjell Axelsson, Prof, University Hospital Orebro, Orebro, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAK-total
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Last update posted 2008-11-27 (Estimated); Status verified 2008-11

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Local infiltration analgesia; Knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Ketorolac; Epinephrine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Group A(Active) (Active Comparator): Group A (Active) receives a multimodal injection intra- and postoperatively
  Interventions: Drug: ropivacaine, ketorolac and epinephrine
- 2 Group P (Placebo) (Placebo Comparator): Group P (Placebo) receives no injection intraoperatively and a saline injection postoperatively
  Interventions: Drug: saline

INTERVENTIONS:
Drug: ropivacaine, ketorolac and epinephrine — In Group A, 400 mg ropivicaine, 30 mg ketorolac and 0.5 mg epinephrine (total volume 166 ml) are infiltrated by the surgeon into the soft tissues peri-articularly during the operation in the following way: Before inserting the components, 20-30 ml are injected into the posterior capsule and before closure of the wound the rest is injected into the capsule incision, the synovium, the ligament and the subcutaneous tissue. After 21 postoperative hours in Group A, 200 mg ropivicaine, 30 mg ketorolac and 0.1 mg epinephrine, total volume 22 ml, are injected intraarticularly via the catheter.
  Arms: 1 Group A(Active)
Drug: saline — In Group P (placebo) no injections were given intraoperatively. All patients had a tunnelled intra-articular multihole 20-G catheter placed at the end of the operation by the surgeon.After 21 postoperative hours 22 ml of saline was injected intraarticularly via the catheter.
  Arms: 2 Group P (Placebo)

SUMMARY:
The primary aim of this study is to evaluate if intra- and postoperative administration of ropivacaine, ketorolac and epinephrine into the operating field would affect morphine consumption. Secondary end-points are hospital stay, pain intensity and side effects. In an attempt to assess the safety of this technique, knee function and patient satisfaction scores are assessed up to 3 months after surgery.

DETAILED DESCRIPTION:
Postoperative pain is often severe following knee arthroplasty. Recently, a local infiltration analgesia (LIA) technique was developed by Drs Kerr and Kohan in Sydney, Australia. With this LIA-technique, a long-acting local anesthetic (ropivacaine), a nonsteroidal anti-inflammatory drug (ketorolac), and epinephrine are infiltrated intraoperatively and via an intraarticular catheter postoperatively. We ahve completed a study on unicompartmental knee arthroplasty and the present study is investigating total knee arthroplasties.

The primary aim of this study is to evaluate if intra- and postoperative administration of ropivacaine, ketorolac and epinephrine into the operating field would affect morphine consumption. Secondary end-points are hospital stay, pain intensity and side effects. In an attempt to assess the safety of this technique, knee function and patient satisfaction scores are assessed up to 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for total knee arthroplasty
* Aged 20-85 yrs
* ASA physical status I-III and mobility indicating normal postoperative mobilization

Exclusion Criteria:

* Known allergy or intolerance to one of the study drugs
* Serious liver-, heart- or renal decease
* Rheumatoid arthritis
* Chronic pain or bleeding disorder

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-04; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 0-48 hours

SECONDARY OUTCOMES:
hospital stay, pain intensity, side effects, knee function and patient satisfaction scores | 0-3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Axelsson, Prof, Principal Investigator — University Hospital Orebro, Sweden
Locations (1):
- University Hospital Orebro, Örebro, Sweden